CLINICAL TRIAL: NCT06977464
Title: Application and Benefit Evaluation of Wearable Technology and Information Software-Based Psychological Stress Monitoring in Return-to-Work Healthcare for Injured Workers: A Longitudinal Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202503083RIND
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Injury; Return to Work; Mental Health
MeSH Terms: conditions — Wounds and Injuries; Psychological Well-Being | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable Technology and Information Software-Based Psychological Stress Monitoring (Active Comparator): The intervention group will additionally use a smartwatch for physiological monitoring and a mobile app for daily to weekly psychological assessments.
  Interventions: Device: Wearable Technology and Information Software-Based Psychological Stress Monitoring
- Control (No Intervention): All participants will receive standard outpatient care.

INTERVENTIONS:
Device: Wearable Technology and Information Software-Based Psychological Stress Monitoring — The intervention group will additionally use a smartwatch for physiological monitoring and a mobile app for daily to weekly psychological assessments.
  Arms: Wearable Technology and Information Software-Based Psychological Stress Monitoring

SUMMARY:
Objective This study aims to develop and evaluate a multidisciplinary service model that integrates wearable devices and mobile health applications to monitor the physical and mental health of workers with occupational injuries during their return-to-work process.

Background With advances in digital health, smartwatches and mobile applications are increasingly used in healthcare to support personalized monitoring and intervention. This project targets injured workers attending occupational medicine clinics, using smartwatches to monitor physiological data and a mobile application to assess psychological status. The model includes remote mental health support and aims to assess its impact on return-to-work outcomes and psychological well-being.

Methods A total of 120 eligible injured workers will be randomly assigned to an intervention or control group. All participants will receive standard outpatient care. The intervention group will additionally use a smartwatch for physiological monitoring and a mobile app for daily to weekly psychological assessments. The 6-month follow-up will evaluate return-to-work success rate, time to return, post-return quality of life, and mental health status.

Intervention Tools The NTU Medical Genie, Labfront, and LINE@ platforms will facilitate real-time monitoring and batch downloading of smartwatch data, as well as the distribution of mood and stress-related questionnaires. At least three occupational rehabilitation education modules will be developed, and case managers will deliver individualized health education and psychological support.

Expected Outcomes The study will assess the effectiveness of this technology-supported, cross-disciplinary care model in improving return-to-work outcomes, mental health, and quality of life. It will also explore participant satisfaction and acceptance of the model. The findings are expected to inform future occupational health interventions and enhance care quality for injured workers.

ELIGIBILITY:
Inclusion Criteria:

* (1) Injured workers aged 18 to 65 years.
* (2) Currently receiving follow-up care at the occupational medicine outpatient clinic of this hospital.
* (3) Expressed willingness to return to work.
* (4) Ability to access the internet and operate the mobile application using a smartphone.

Exclusion Criteria:

* (1) Individuals not expected to regain work capacity of at least 3 hours per day within six months.
* (2) Individuals who have resigned and do not intend to return to work within six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Return to work | 6 months
  Successful return to work (defined as resumption of work with fewer than six weeks of subsequent sick leave) and the duration from initial clinic visit to return to work.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided